CLINICAL TRIAL: NCT03708367
Title: A Post-Market Evaluation of LipiFlow Treatment in Cataract Surgery Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DRYE-102-SELF
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Cataracts; Meibomian Gland Dysfunction (MGD)
MeSH Terms: conditions — Cataract; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Group: LipiFlow Treatment at PreOp (Experimental): Study subjects that meet all inclusion and exclusion criteria will be randomized to receive LipiFlow Thermal Pulsation System treatment at preoperative visit before bilateral implantation with commercially-available Symfony Intraocular Lens
  Interventions: Device: LipiFlow Thermal Pulsation System
- Control Group (Other): Study subjects that meet all inclusion and exclusion criteria will be randomized to not receive the LipiFlow Thermal Pulsation System treatment at a preoperative visit before bilaterally implanted with the commercially available Symfony Intraocular Lens. Control Group will receive LipiFlow treatment as cross-over group at 3 months postoperative visit.
  Interventions: Device: LipiFlow Thermal Pulsation System

INTERVENTIONS:
Device: LipiFlow Thermal Pulsation System — Treatment at preoperative visit for study group
  Arms: Study Group: LipiFlow Treatment at PreOp
Device: LipiFlow Thermal Pulsation System — Treatment at 3 month visit as the cross-over group
  Arms: Control Group

SUMMARY:
This is a post-market, prospective, randomized, multi-center, bilateral, open-label, cross-over, comparative clinical study. Study group will undergo preoperative LipiFlow treatment and Control group will not receive preoperative LipiFlow treatment. Three months postoperatively, both groups will be evaluated for clinical outcomes and the Control group will receive LipiFlow treatment as the cross-over group. The Control group will be evaluated at 4 months postoperative for clinical outcomes.

ELIGIBILITY:
Inclusion Criteria (all criteria apply to each study eye):

* Minimum 22 years of age.
* Bilateral cataracts for which phacoemulsification extraction and implantation with Symfony IOLs have been planned.
* Evidence of Meibomian Gland Dysfunction (MGD) in both eyes based on assessment of meibomian glands of the lower eyelid
* None to moderate dry eye symptoms with questionnaire
* Clear intraocular media other than cataract in each eye.
* Availability, willingness, ability and sufficient cognitive awareness to comply with the study protocol including: randomization; examination procedures; completion of planned bilateral cataract surgeries; compliance with no use of other MGD or dry eye treatments.
* Ability to understand, read and write English to consent to study participation and complete study questionnaires.
* Willingness to sign informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing country.

Exclusion Criteria (all criteria apply to each study eye):

* Any medical finding that would predictably result in a postoperative best corrected distance visual acuity worse than 20/30 in either eye.
* Use of systemic or ocular medications that, in the opinion of the investigator, may affect vision or impact pupil dilation or iris structure.
* Irregular corneal astigmatism.
* Any clinically-significant corneal pathology / abnormality other than regular corneal astigmatism.
* Any clinically-significant pupil abnormalities.
* Subjects with conditions associated with increased risk of zonular rupture.
* Unwillingness or inability to stop wearing contact lens at least two weeks prior to the baseline visit.
* Known ocular disease or pathology that, in the opinion of the investigator, may affect visual acuity or require surgical intervention during the study.
* Systemic disease condition that causes dry eye.
* Unwillingness or inability to abstain from the use of systemic medications known to cause dryness for the study duration. Subjects must have discontinued these medications for at least 1 month prior to Preoperative Visit.
* Unwillingness or inability to abstain from the use of systemic antihistamines.
* Unwillingness or inability to abstain from use of prescription medications for treatment of MGD or dry eye. Subject must have dicontinued using prescription medications for MGD or dry eye at least 1 month prior to baseline preoperative visit #1 measurements.
* Any of the following ocular (eye or eyelid) conditions in either eye within 3 months prior to the LipiFlow treatment visit:

  * Prior intraocular, oculoplastic, corneal or refractive surgery procedure (LASIK, LASEK, RK, PRK, etc.).
  * Ocular trauma.
  * Ocular Herpes simplex or Herpes zoster (eye or eyelid) infection.
  * History of recurrent ocular inflammation.
  * Punctal plug insertion or punctal occlusion.
* Any of the following active ocular (eye or eyelid) conditions in either eye at the baseline Preoperative Visit #1 measurements:

  * Ocular infection.
  * Ocular inflammation.
  * Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis
  * Severe (Grade 3 or 4) inflammation of the eyelid.
  * Eyelid abnormalities that affect lid function.
  * Ocular surface abnormality that may compromise corneal integrity.
* Concurrent participation or participation within 30 days prior to study visit in any other clinical trial.
* Planned monovision correction.
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Janakiraman, OD, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (5):
- United States (5):
  - Empire Eye & Laser Center, Inc., Bakersfield, California
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Matossian Eye Associates, Pennington, New Jersey
  - JW Eye Associates, P.A., Dallas, Texas
  - Texas Eye & Laser Center, P.A., Hurst, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matossian C, Chang DH, Whitman J, Clinch TE, Hu J, Ji L, Murakami D, Wang Y, Blackie CA. Preoperative Treatment of Meibomian Gland Dysfunction with a Vectored Thermal Pulsation System Prior to Extended Depth of Focus IOL Implantation. Ophthalmol Ther. 2023 Oct;12(5):2427-2439. doi: 10.1007/s40123-023-00740-x. Epub 2023 Jun 15. PMID 37318707

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All study subjects enrolled from the normal surgical cataract population with bilateral mild to moderate Meibomian Gland Dysfunction, scheduled for bilateral cataract surgeries with Symfony Intraocular Lens implantation, at 5 sites in the U.S.A. 143 Subjects were consented, 26 screen-failed and 117 were randomized and bilaterally implanted. 115 evaluable subjects completed the study (58 in the study group and 57 in the Control Group).
Units Other Than Participants: Eyes
Groups:
- Study Group: LipiFlow treatment at Pre-operative
- Control Group: LipiFlow treatment following 3-month visit
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 59; 117 Eyes | 58; 115 Eyes
Completed | 58; 116 Eyes | 57; 114 Eyes
Not Completed | 1; 1 Eyes | 1; 1 Eyes

BASELINE CHARACTERISTICS:
Population: All eyes that are randomized and implanted
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 59 | 58 | 117
Number analyzed (Eyes) | 117 | 115 | 232
Age, Customized [Number; unit: Participants]
  30-39 years | 1 | 0 | 1
  40-49 years | 1 | 1 | 2
  50-59 years | 13 | 10 | 23
  60-69 years | 28 | 31 | 59
  >=70 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 57 | 55 | 112
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (Including Indian) | 3 | 4 | 7
  Black | 8 | 12 | 20
  Caucasian | 48 | 42 | 90

OUTCOME MEASURES:

1. Primary Outcome: Mean Monocular UCDVA (Uncorrected Distance Visual Acuity)
Description: Uncorrected Distance Visual Acuity was measured for the Study and Control groups at the 3-month visit using the Clinical Trial Suite (M&S Technologies) at 4.0 meters under photopic conditions (~85 cd/m2).
Time Frame: 3 months Postoperative
Population: Results from both eyes from all randomized subjects were included. Not all subjects completed all tests.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 58 | 57
Number analyzed (Eyes) | 116 | 114
LogMAR | 0.08 (0.15) | 0.07 (0.13)

2. Primary Outcome: Precision (Standard Deviation) of Preoperative Keratometric Measurements
Description: Biometry testing was done pre-operatively
Time Frame: 2-4 weeks after first Pre-operative visit
Population: Results from both eyes from all randomized subjects were included. Not all subjects completed all tests.
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: Eyes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 56 | 58
Number analyzed (Eyes) | 112 | 116
diopter
  Precision of Keratometry 1 (K1) | 0.0 (0.09) | -0.01 (0.07)
  Precision of Keratometry 2 (K2) | 0.0 (0.09) | 0.0 (0.07)

3. Primary Outcome: Precision of Axial Length (AL) and Anterior Chamber Depth (ACD)
Description: Biometry testing was done pre-operatively
Time Frame: 2-4 weeks after first Pre-operative visit
Population: Results from both eyes from all randomized subjects were included. Not all subjects completed all tests.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 56 | 58
Number analyzed (Eyes) | 112 | 116
mm
  Precision of Axial Length (AL) | 0.0 (0.02) | 0.0 (0.01)
  Precision of Anterior Chamber Depth (ACD) | 0.0 (0.01) | 0.0 (0.02)

4. Primary Outcome: Rate of Refractive Predictability
Description: Percentage of eyes with achieved manifest refractive spherical equivalence (MRSE) within +/- 0.50 D and +/- 1.00 D.
  Achieved MRSE for each eye is defined as postoperative MRSE minus targeted MRSE.
Time Frame: Difference between Baseline visit and Postoperative visit at 10-14 weeks after cataract surgery on the second eye.
Population: Results from both eyes from all randomized subjects were included. Not all subjects completed all tests.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 58 | 57
Number analyzed (Eyes) | 116 | 114
Percentage of eyes
  +/- 0.50 D | 73.3 | 82.5
  +/- 1.00 D | 94.0 | 98.2

5. Primary Outcome: Rate of Bothersome Ocular Symptoms
Description: Patient-Reported Visual Symptom Questionnaire (PRVSQ) Rating Results at 3 months postoperative
Time Frame: 3 months postoperative
Population: Questionnaires were completed by bilaterally implanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 58 | 57
Participants
  Q1a) Halos over the last 7 days | 34 | 45
  Q2a) Starburst over the last 7 days | 36 | 40
  Q3a) Multiple or Double vision over the last 7 days | 15 | 5
  Q4a) Sensitivity to Light over the last 7 days | 38 | 33
  Q5a) Glare related to scattered light over the last 7 days | 20 | 28
  Q6a) Occlusions over the last 7 days | 1 | 2
  Q7a) Poor Low Light Vision over the last 7 days | 36 | 33

6. Primary Outcome: Mean Change in Total Meibomian Gland Score From Baseline to 1 Month Postoperative
Description: Total Meibomian Gland Score: Fifteen Meibomian Glands (five temporally, centrally and nasally) in the lower eye are assessed on a scale of 0 - 3 (0 - No secretion, 1 - Inspissated (toothpaste consistency), 2 - Colored/cloudy liquid secretion or 3 - Clear liquid oil secretion). The sum of all 15 glands constitute the total meibomian gland secretion score (range 0-45).
Time Frame: Preoperative Visit (Baseline) and Postoperative Visit between 30-60 days after cataract surgery on the second eye.
Population: Results from both eyes from all randomized subjects were included. Not all subjects completed all tests.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 57 | 57
Number analyzed (Eyes) | 114 | 114
Units on a scale | 4.8 (8.2) | 3.9 (8.3)

ADVERSE EVENTS:
Time Frame: 3 months for study group and 4 months for available control group
Groups:
- Control Group: Prior to LipiFlow treatment at 3-month visit
- Control Group: AEs occurring after LipiFlow treatment
Arm/Group | Study Group | Control Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58 | 0/56
Serious Adverse Events (participants affected / at risk) | 3/59 | 4/58 | 1/56
Other Adverse Events (participants affected / at risk) | 0/59 | 2/58 | 5/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=59) | Control Group (N=58) | Control Group (N=56)
Anterior Capsular Phimosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cystoid Macular Edema (Eye disorders) | 1 (1) | 2 (3) | 0 (0)
Hospitalization - Neck procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hospitalization- fall related to dehydration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hospitalization- shingles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hospitalization-ischemic event (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=59) | Control Group (N=58) | Control Group (N=56)
Undesirable Optical Phenomena (Surgical and medical procedures) | 0 (0) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (2):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03708367/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT03708367/SAP_001.pdf